CLINICAL TRIAL: NCT05655923
Title: Clinical and Biochemical Assessment of Ozonated Olive Oil Mixed Bone Substitute in Treating Intra Bony Periodontal Defect- Randomized Clinical Trial
Brief Title: Clinical and Biochemical Assessment of Ozonated Olive Oil Mixed Bone Substitute in Treating Intra Bony Periodontal Defect
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nourhan adel mohammed mahmoud aldorri, doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ozonized oil in periodontitis
Record Dates: First submitted 2022-12-10; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Periodontitis
Keywords: intrabony defect
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: ozonized olive oil
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Placebo Comparator): ten patients will be subjected to place bone substitute mixed with Olive oil in intra bony defect. ( Control group)
  Interventions: Biological: xenograft bone substitute
- Group II (Active Comparator): ten patients will be subjected to place bone substitute mixed with ozonated olive oil in intra bony defect without further application of ozonated oil.
  Interventions: Biological: ozonized olive oil; Biological: xenograft bone substitute
- Group III (Active Comparator): ten patients will be subjected to place bone substitute mixed with ozonated olive oil in intra bony defect with further weekly application of ozonated olive oil until third week
  Interventions: Biological: ozonized olive oil; Biological: xenograft bone substitute

INTERVENTIONS:
Biological: ozonized olive oil — ozonized oil will be mixed with xenograft in group II and Group III
  Arms: Group II; Group III
Biological: xenograft bone substitute — Xenograft bone substitutes in all Groups
  Other Names: deproteinized bovine bone

SUMMARY:
The goal of this study is to investigate the effect of ozonated olive oil in treating intra bony defect by means of clinical and radiographic parameters, and gingival cervicular fluid BMP2 level.

DETAILED DESCRIPTION:
Ozone is a triatomic molecule, containing three oxygen atoms. has many different uses in various fields; one of them is a practice of ozone in medicine (Seidler et al, 2008) as well as in dentistry field(Azarpazhooh & Limeback 2008). Ozone is unstable gas and release rapidly a nascent oxygen molecule to form an oxygen gas, due to this property ozone gas used to kill bacteria, fungi, Inactivate viruses, and control bleeding.(Gupta & Mansi, 2012).

There are three different systems for producing ozone gas: Ultraviolet System: yields low concentrations of ozone, used in, saunas, esthetics and for air decontamination. Cold Plasma System: used in water and air decontamination. Corona Discharge System yields a high amount of ozone. Most commonly used system, corona discharge system easy to manipulate and has a precise ozone production amount. (Gupta & Mansi, 2012). Ozone has three forms of application in dentistry ozonated water, ozonated olive oil, ozone gas. Ozonated olive oil and water show an ideal system to be used due to the ability to trap and discharges oxygen /ozone. (Meena et al, 2011).

The aims of oxygen/ozone therapy are removal of pathogens, reestablishment of proper oxygen metabolic rate, stimulation of a pleasant ecologic environment, improve circulation, immune stimulation, stimulation of an anti-oxidant system.(Gattani & Shewale, 2016).

antimicrobial (antibacterial, antifungal, and antiviral) effect is claimed to be through damaging to the cytoplasmic membrane, oxidation of intracellular content specific to the microbial cell, effective in antibiotic resistive strain. Nagayoshi M et al 2004 conducted a study to evaluate the ability of different concentrations of ozone on survival and permeability of oral microorganisms. they reported that ozonated water (0.5-4 mg/l) was greatly effective in killing both gram-positive and gram-negative bacteria. Some strains of gram-negative bacteria as P. endodontalis and the periodontopathic bacterium P. gingivalis shows more liability to ozonated water than gram-positive bacteria.(Nagayoshi et al, 2004). Immunostimulate effect of ozone therapy was reported to be related to its effect on triggering cellular and humoral immune system, Proliferation of immunocompetent cells, Synthesis of immunoglobulin's, Enhance phagocytosis activity (V. Bocci, n.d.). Ozone therapy was found also to have an active role in activation of antioxidants and synthesis of interleukin, leukotriene, and prostaglandin.( V. Bocci et al, 2009, Gattani & Shewale, 2016) A systematic review by (V. A. Bocci et al, 2011) was conducted to study the interaction of ozone therapy and blood. In erythrocytes, it activates phosphofructokinase, thus accelerate glycolysis and result in increased ATP and 2, 3-diphosphoglycerate. Repeated sessions, allow lipid oxidation products to reach bone marrow and activate subtle development at erythropoietin level, this will form new erythrocytes and improved its biochemical characteristics, a phenomena named "super gifted erythrocytes". This super gifted erythrocytes was found to have a high content of glucose-6-phosphate dehydrogenase. Ozone therapy enhanced the phagocytosis effect of neutrophil and trigger cysteine oxidation and induce the release of cytokines. During the ozone therapy, detection of platelet-derived growth factor, subunit B, TGF-b1, IL- 8 and epidermal growth factor released in heparinized plasma(Bocci et al, 2011). A recent randomized controlled trial was conducted to study the efficiency of ozone therapy in an early healing period of connective tissue gingival graft placed to cover root surface (Taşdemir et al. 2016)they concluded that, ozone therapy improved blood profusion during the first week of therapy which could improve wound healing and decrease post-operative pain.

(Patel et al, 2011) evaluated the therapeutic effects of topical ozonized olive oil on the healing of post-harvested palatal donor wound sites, with large epithelial and connective tissue deficiencies that heal by secondary intention. The result revealed that ozonized oil significantly enhanced re-epithelialization of the palatal donor site wounds.

The main challenge facing periodontal therapy is that of contamination during the early phases of healing which compromise the initial healing events. In addition, the tissue response to such inflammatory state that usually associated with marked reduction in anabolic mediators also compromise periodontal regeneration. Since ozone therapy works on both bacterial, inflammatory and host anabolic and catabolic mediators, it should be studied carefully in order to investigate more and augment its role in periodontal therapy.We still have few investigations with lots of gaps still needs to be investigated. Thus this study will be performed to approach the effect of ozonized olive oil mixed with the bone substitute as a biocompatible scaffold and as a possible delivery material in treating Intra-bony periodontal defects.

ELIGIBILITY:
Inclusion Criteria:

chronic periodontitis requiring surgical intervention to treat an intra-bony defect adjacent to a natural tooth One or more periodontal defects with PD >6 mm, radiographic vertical bony defect >3 mm in depth, and radiographic base of defect >2 mm coronal to the root apex.

Systemically healthy as evidence by a medical questionnaire guided by modified cornel medical index Availability for multiple follow-up appointments.

Exclusion Criteria:

Smokers women who were pregnant or intended to become pregnant during the study period Patient unwilling to perform hygienic instructions Untreated infection at the study site other than periodontitis Tooth mobility Miller Class II or III Subgingival restoration, untreated caries at or below the cement enamel junction (CEJ), root fracture, or apical pathology.

Vulnerable individuals Presence of systemic diseases.

-

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
intrabony defect fill | 6 months
  regeneration of intrabony defect with enhance in clinical parameter

SECONDARY OUTCOMES:
BMP2 | 3 weeks
  increase of GCF of bone morphogenic protein 2

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azarpazhooh A, Limeback H. The application of ozone in dentistry: a systematic review of literature. J Dent. 2008 Feb;36(2):104-16. doi: 10.1016/j.jdent.2007.11.008. Epub 2007 Dec 31. PMID 18166260
- [Background] Bocci VA, Zanardi I, Travagli V. Ozone acting on human blood yields a hormetic dose-response relationship. J Transl Med. 2011 May 17;9:66. doi: 10.1186/1479-5876-9-66. PMID 21575276
- [Background] Nagayoshi M, Fukuizumi T, Kitamura C, Yano J, Terashita M, Nishihara T. Efficacy of ozone on survival and permeability of oral microorganisms. Oral Microbiol Immunol. 2004 Aug;19(4):240-6. doi: 10.1111/j.1399-302X.2004.00146.x. PMID 15209994
- [Background] Laurell L, Gottlow J, Zybutz M, Persson R. Treatment of intrabony defects by different surgical procedures. A literature review. J Periodontol. 1998 Mar;69(3):303-13. doi: 10.1902/jop.1998.69.3.303. PMID 9579616
- [Background] Patel PV, Kumar V, Kumar S, Gd V, Patel A. Therapeutic effect of topical ozonated oil on the epithelial healing of palatal wound sites: a planimetrical and cytological study. J Investig Clin Dent. 2011 Nov;2(4):248-58. doi: 10.1111/j.2041-1626.2011.00072.x. Epub 2011 Jul 7. PMID 25426896
- [Background] Tasdemir Z, Alkan BA, Albayrak H. Effects of Ozone Therapy on the Early Healing Period of Deepithelialized Gingival Grafts: A Randomized Placebo-Controlled Clinical Trial. J Periodontol. 2016 Jun;87(6):663-71. doi: 10.1902/jop.2016.150217. Epub 2016 Jan 16. PMID 26777769